CLINICAL TRIAL: NCT00766753
Title: A Phase I/II Evaluation of Vaccination With Type 1 Dendritic Cells Pulsed With Multiple Peptides in the Treatment of HLA-A2 Positive Patients With Recurrent Malignant Gliomas
Brief Title: Vaccination-Dendritic Cells With Peptides for Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Frank Lieberman (Other)
Collaborators: Oncovir, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Frank Lieberman, Professor of Neurology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-115; NIH/NINDS/NCI; 1R21CA117152-01A2 (NIH)
Record Dates: First submitted 2008-06-23; First posted 2008-10-06 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Malignant Glioma
Keywords: HLA-A2 positive; Malignant Gliomas; Vaccine
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single (Experimental): All consenting, eligible subjects receive the intervention
  Interventions: Biological: Dendritic vaccine pulsed with multiple peptides; Biological: The first booster vaccine phase:; Biological: The second booster vaccine phase:

INTERVENTIONS:
Biological: Dendritic vaccine pulsed with multiple peptides — Subjects will receive four (4) injections of the vaccine into the lymph nodes. Injection is guided by ultrasonography. Subjects will receive the first cycle of vaccine in the right groin. Two weeks after the first vaccine, subjects receive the same vaccine at the left groin, followed by the 3rd and the 4th vaccines in the left and right armpits, respectively, with two-week intervals. Each injection contains 0.2cc (less than 1/20th of a teaspoon) of a saline solution containing the vaccine cell mixture.
Biological: The first booster vaccine phase: — This phase will begin at week 13. These subjects will be treated with additional vaccinations every 4 weeks to a maximum of 5 vaccine injections and, if poly-ICLC is available from the supplier starting on the day of the first additional vaccine and twice/week for 8 injections following each additional vaccine. If poly-ICLC supply is not available from the supplier, DC vaccines only will be given in the booster phases.
Biological: The second booster vaccine phase: — At week 33, following the completion of 5 additional vaccines, if participants demonstrate stable disease or positive clinical response, if poly-ICLC supply is still available, participants will be offered additional DC-vaccines and poly-ICLC treatment. The second phase booster vaccines can be continued as long as the patient shows continued positive response or stable disease (both radiological and clinically) with no major adverse events, and as long as funding is available for the study. DC vaccines in this phase will be administered every 6 months+/- 2 weeks.
  2). Poly-ICLC at 10µg/kg and up to 1640 µg/injection will be administered intramuscularly (i.m.) on the day of each booster DC vaccine. Poly-ICLC will be administered weekly thereafter for twice (at one week and two weeks after each vaccine) (e.g. if the previous DC vaccine was administered on a Thursday, subsequent poly-ICLC will be administered on the next two Thursdays

SUMMARY:
This is a single-institution Phase I/II study designed to evaluate the safety and induction of an immune response, and preliminary clinical response of vaccinations with Type-1 alpha-DCs (alpha-DC1) loaded with glioma-associated antigen (GAA) epitopes and administration of poly-ICLC in patients with recurrent malignant gliomas. Approximately 30 subjects will be enrolled in this study at UPMC/UPCI Hillman Cancer Center. The study participants in this trial will be HLA-A2 positive male or female adults over 18 years of age. The primary objective is to establish the safety of this approach. The endpoints will be to determine the maximum tolerated dose (MTD) of alpha-DC1 vaccines in combination with a fixed dose of poly-ICLC, using standard criteria and close clinical followups. The secondary objectives are 1) to assess the immunological response against GAAs in patients with recurrent malignant gliomas immunized with DCs loaded with GAA-derived peptides using enzyme-linked immuno-spot (ELISPOT), delayed-type hypersensitivity (DTH) and tetramer assays; and 2) to assess the preliminary anti-tumor clinical activity of the vaccines as measured by radiological response (MRI), overall survival, and 4- and 6-month progression-free survival (PFS).

DETAILED DESCRIPTION:
This is a single-institution Phase I/II study designed to evaluate the safety, the induction of an immune response, and the preliminary clinical response of vaccinations with Type-1 αDCs (αDC1) loaded with glioma-associated antigen (GAA) epitopes and administration of poly-ICLC in patients with recurrent malignant gliomas. The hypothesis is that this form of vaccines in combination with poly-ICLC treatment will prove to be safe, and will induce potent anti-glioma immune responses.

The primary objective is to establish the safety of the approach.

The secondary objectives are to 1) assess the immunological response against GAAs in patients with recurrent malignant gliomas immunized with DCs loaded with GAA-derived peptides using enzyme-linked immuno-spot (ELISPOT), delayed-type hypersensitivity (DTH) and tetramer assays and 2) assess the preliminary anti-tumor clinical activity of the vaccines as measured by radiological response (MRI), overall survival, and four- and six-month progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed

  * recurrent glioblastoma (GBM)
  * anaplastic astrocytoma (AA)
  * anaplastic oligodendroglioma (AO)
  * anaplastic mixed oligoastrocytoma (AMO)
  * other anaplastic glioma
* Patients must have received prior external beam radiotherapy and/or chemotherapy unless patients refused the options.
* Patients may have had treatment for no more than 2 prior relapses. Relapse is defined as progression following initial therapy (i.e. radiation +/- chemo if that was used as initial therapy).
* Patients must be HLA-A2 positive.
* All patients must sign an informed consent document indicating that they are aware of the investigational nature of this study.
* Patients must sign an authorization for the release of their protected health information.
* Patients must be > 18 years old, and with a life expectancy > 8 weeks. -Patients must have a Karnofsky performance status of > 60.
* Patients must have recovered from the toxic effects of prior therapy: 4 weeks from any investigational agent, 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 4 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the principal investigator.
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism.
* Patients must not have any serious concurrent medical illness.
* Documented negative serum beta-HCG for female patients of child-bearing age.
* Patients must be free of systemic infection. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment.
* Patients must have adequate organ function as measured by:

  1. Hematopoietic:

     * granulocytes at least 2500/mm3
     * lymphocytes at least 1000/mm3
     * platelets at least 100,000/mm3
     * hemoglobin at least 10.0 g/dL
  2. Cardiac: Asymptomatic or, if symptomatic, then left ventricular ejection fraction at rest must be at least 50% or within the normal range of the institution. A cardiology clearance will be required for LV ejection fraction 50%.
  3. Hepatic: AST, ALT, GGT, LDH, Alk phos within 2.5 x upper normal limit and total bilirubin no greater than 2.0 mg/dL.
  4. Renal: Serum creatinine up to 1.5 x upper normal limit.
  5. Pretreatment baseline evaluations for laboratory parameters must be obtained within 10 to 18 days of subject registration.

Exclusion Criteria:

* Pregnant or breast-feeding.
* Presence of metastatic disease.
* Active bacterial, viral or fungal infections. Subjects with active infections (whether or not they require antibiotic therapy) may be eligible after complete resolution of the infection. Subjects on antibiotic therapy must be off antibiotics for at least 7 days before beginning treatment.
* Chemotherapy, biologic therapy or radiation therapy less than one month prior to study entry.
* History or presence of autoimmune disease.
* Use of immunosuppressives within 4 weeks prior to study entry or anticipated use of immunosuppressive agents. Minimum doses of corticosteroid (dexamethasone up to 4 mg/day) is permitted.
* Subjects with uncontrolled pain. -Subjects who have sensitivity to drugs to provide local anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-12 (Actual); Primary Completion 2009-09 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Lieberman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Online database of trials; this links the viewer to the UPMC website — http://www.virtualtrials.com/vaccine.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- AlphaDC1 - Dose Level 1(1 X 10 7) + Poly-ICLC; AlphaDC1 - Dose Level 2 (3 x 10 7) + Poly-ICLC: Patients with recurrent malignant glioma treated with novel vaccination with -type 1 polarized dendritic cells ( DC1) loaded with synthetic peptides for glioma-associated antigen (GAA) epitopes and administration of polyinosinic-polycytidylic acid [poly(I:C)] stabilized by lysine and arboxymethylcellulose (poly-ICLC)
Period: Overall Study
Arm/Group | AlphaDC1 - Dose Level 1(1 X 10 7) + Poly-ICLC | AlphaDC1 - Dose Level 2 (3 x 10 7) + Poly-ICLC
Started | 11 | 11
Received at Least One Vaccine | 11 | 11
Completed at Least Four Vaccines | 10 | 9
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with recurrent malignant glioma treated with novel vaccination with type 1 polarized dendritic cells ( DC1) loaded with synthetic peptides for (GAA) epitopes and administration of polyinosinic-polycytidylic acid [poly(I:C)] stabilized by lysine and arboxymethylcellulose (poly-ICLC) who received at least one vaccine up to 4 vaccines
Groups:
- Total: Total of all reporting groups
Arm/Group | AlphaDC1 - Dose Level 1(1 X 10 7) + Poly-ICLC | AlphaDC1 - Dose Level 2 (3 x 10 7) + Poly-ICLC | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Median (Full Range); unit: years] | 52 [37 to 71] | 46 [28 to 63] | 48 [28 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-related Dose Limiting Toxicities (DLT)
Description: Number of participants who experienced treatment-related Dose Limiting Toxicities (DLT) at any dose level.
Time Frame: up to 8 weeks
Population: Participants at any dose level, through the first booster phase.
Measure: Count of Participants; unit: Participants
Groups:
- AlphaDC1 - Dose Level 1(1 X 10^7) + Poly-ICLC; AlphaDC1 - Dose Level 2 (3 x 10^7) + Poly-ICLC: Patients with recurrent malignant glioma treated with novel vaccination with -type 1 polarized dendritic cells ( DC1) loaded with synthetic peptides for glioma-associated antigen (GAA) epitopes and administration of polyinosinic-polycytidylic acid [poly(I:C)] stabilized by lysine and arboxymethylcellulose (poly-ICLC)
Arm/Group | AlphaDC1 - Dose Level 1(1 X 10^7) + Poly-ICLC | AlphaDC1 - Dose Level 2 (3 x 10^7) + Poly-ICLC
Number analyzed (Participants) | 11 | 11
Participants | 0 | 0

2. Primary Outcome: Median Time To Progression
Description: Median number of months until disease progression. Tumor size was assessed using magnetic resonance imaging (MRI) scans with contrast enhancement to detect change from baseline.
Time Frame: At baseline, 9, 17, 25, and 33 weeks, and every 3 months; up to 23 months
Population: as for baseline characteristics
Measure: Median (Full Range); unit: months
Arm/Group | AlphaDC1 - Dose Level 1(1 X 10 7) + Poly-ICLC | AlphaDC1 - Dose Level 2 (3 x 10 7) + Poly-ICLC
Number analyzed (Participants) | 11 | 11
months
  WHO3 AG (anaplastic glioma) | 5 [0 to 23] | 15 [0 to 23]
  WHO4 GBM (glioblastoma multiforme) | 4 [0 to 23] | 4 [0 to 23]

3. Secondary Outcome: 12-month- Progression Free Survival (PFS)
Description: Number of patients with progression-free status lasting at least 12 months
Time Frame: Up to 12 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | AlphaDC1 - Dose Level 1(1 X 10 7) + Poly-ICLC | AlphaDC1 - Dose Level 2 (3 x 10 7) + Poly-ICLC
Number analyzed (Participants) | 11 | 11
participants
  AA (anaplastic astrocytoma) | 2 | 1
  AO (anaplastic oligodendroglioma) | 1 | 1
  AOA (anaplastic oligoastrocytoma) | 0 | 1
  GBM (glioblastoma multiforme) | 2 | 2

4. Secondary Outcome: Overall Survival (OS)
Description: Time interval from start of treatment until date of death.
Time Frame: Up to 102 months
Population: as for baseline characteristics
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | AlphaDC1 - Dose Level 1(1 X 10^7) + Poly-ICLC | AlphaDC1 - Dose Level 2 (3 x 10^7) + Poly-ICLC
Number analyzed (Participants) | 11 | 11
months | 32.88 [13.58 to 36.59] | 13.28 [5.59 to 36.79]

ADVERSE EVENTS:
Groups:
- Alpha DC1 Vaccine + Poly-ICLC: Patients with recurrent malignant glioma treated with novel vaccination with -type 1 polarized dendritic cells ( DC1) loaded with synthetic peptides for (GAA) epitopes and administration of polyinosinic-polycytidylic acid [poly(I:C)] stabilized by lysine and arboxymethylcellulose (poly-ICLC) who received at least one vaccine, up to 4 vaccines
Arm/Group | Alpha DC1 Vaccine + Poly-ICLC
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha DC1 Vaccine + Poly-ICLC (N=22)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alpha DC1 Vaccine + Poly-ICLC (N=22)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4
Hypertension (Cardiac disorders) | 2
Weight gain (General disorders) | 2
Insomnia (General disorders) | 4
Rigors/chills (General disorders) | 5
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 7
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 2
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 4
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 13
Diarrhea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Infection with normal ANC or Grade 1 or 2 neutrophils, Sinus (Infections and infestations) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy), Left-sided (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 3
Memory impairment (Nervous system disorders) | 2
Neurology - Other (Specify, __) (Nervous system disorders) | 2
Somnolence/depressed level of consciousness (Nervous system disorders) | 3
Confusion (Nervous system disorders) | 4
Neuropathy: motor (Nervous system disorders) | 4
Seizure (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 5
Neuropathy: sensory (Nervous system disorders) | 5
Pain, Throat/pharynx/larynx (General disorders) | 3
Pain, Muscle (General disorders) | 4
Pain - Other (Specify, __) (General disorders) | 7
Pain, Extremity-limb (General disorders) | 9
Pain, Head/headache (General disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2
Flu-like syndrome (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes